CLINICAL TRIAL: NCT03225885
Title: Effectiveness of Prenatal Counseling for Prematurity Using a Supplementary Multimedia Parent Education Tool
Brief Title: Counseling for Prematurity Using a Multimedia Education Tool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Collaborators: Marquette University (Other); Children's National Research Institute (Other); AMAG Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Mir A Basir, Associate Professor, Medical College of Wisconsin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PRO00028712
Record Dates: First submitted 2017-07-20; First posted 2017-07-21 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Premature Birth; Counseling; Decision Making; Prenatal Care; Infant, Premature; Resuscitation
Keywords: gestational age; multi-media; mobile application; anxiety; clinical trial; random allocation
MeSH Terms: conditions — Premature Birth; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial where participants are assigned to 1 of 2 groups for the duration of the study. One group will receive verbal counseling and a printed gestational age handout. The other group will receive verbal counseling and a bedside iPad with the multimedia information about prematurity.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Printed Handout (Active Comparator): Participants in this arm will receive verbal prematurity counseling from a Neonatologist or Neonatal fellow as well as a printed gestational age specific handout about prematurity.
  Interventions: Other: Printed Handout
- Multimedia Information (Experimental): Participants in this arm will receive verbal prematurity counseling from a Neonatologist or Neonatal fellow as well as have bedside access to iPad multimedia information regarding prematurity.
  Interventions: Other: Multimedia Information

INTERVENTIONS:
Other: Multimedia Information — Is a multi-media mobile application that addresses information about prematurity, resuscitation, and NICU hospitalization.
  Arms: Multimedia Information
Other: Printed Handout — Printed Handout is a gestational age specific handout that addresses resuscitation and prematurity information.
  Arms: Printed Handout

SUMMARY:
This study evaluates the effectiveness of prenatal counseling when verbal counseling is supplemented with a multi-media mobile application versus a written gestational age handout.

DETAILED DESCRIPTION:
Approximately 500,000 infants are born prematurely in the United States every year. Premature birth prior to 27 weeks gestation currently accounts for approximately 40% of infant mortality within the United States. When compared to full term infants, premature infants have a higher risk of physical or cognitive impairment and prematurity care accounts for over 26 billion dollars annually. Parents of premature infants are placed under significant emotional, financial, and personal stress. However, parental education about prematurity is often not evidenced based, varies significantly between OB and Neonatology providers, and lacks educational aids to help parents comprehend the information provided.

Several medical societies (American Academy of Pediatrics (AAP), American Congress of Obstetrics and Gynecology (ACOG), National Institute of Child Health and Human Development (NICHD)) and parental advocates have voiced concern that the current practice is sub-optimal. Several studies have looked at this challenging situation from the family's perspective and have shown that parents find this counseling to be helpful but rarely reassuring and often stressful. Cognitive science research has recommended the use of multimedia information to simultaneously use both text and visual cognitive channels to improve information uptake and retention. Policy statements from the AAP, ACOG, and NICHD have all emphasized the importance of improving the prenatal counseling process to give our parents the most information possible so that they can make the best choices possible for their vulnerable infant.

Potential study participants will be identified after hospitalization at Froedtert Hospital for premature labor. As per current clinical practice all mothers and their support person will have a neonatology consult requested by the obstetrician. These potential participants will be screened for eligibility in the study. Mothers and their support person will then be consented for participation and will be randomized to receive either verbal counseling with printed gestational age handout or verbal counseling with the multimedia information regarding prematurity. Participation of the pregnant woman's support person will be allowed by not required. If both mother and support person consent to participate, the support person will be will be assigned the same group as the mother. Participants will take a baseline STAI (State-Trait Anxiety Inventory) at time of randomization. After prenatal counseling has been completed by a neonatal provider (neonatology attending or fellow) the participants will be provided the validated questionnaire (previously developed) to assess their knowledge of prematurity based on the AAP recommended information for parents anticipating a premature birth. Participants will also retake the STAI.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Admitted to Labor and Delivery unit due to concerns for premature delivery, gestational age of fetus between 22 weeks 0 days and 33 weeks 6 days

Exclusion Criteria:

* known significant genetic abnormality or congenital anomaly that would effect survival or counseling that parents receive
* participants will be excluded from analysis if delivery occurs prior to completion of questionnaires as other sources of information become available after birth

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-01-25 (Actual); Study Completion 2019-01-25 (Actual)

PRIMARY OUTCOMES:
Overall knowledge of prematurity | within 24 hours of verbal counseling session
  Average of overall knowledge score

SECONDARY OUTCOMES:
Gestational age sub-group knowledge scores | within 24 hours of verbal counseling session
  Comparison of average overall knowledge scores within gestational age groups 22-24 weeks and 25-29 weeks and 30-33 weeks gestation.
Sub-domain knowledge scores | within 24 hours of verbal counseling session
  Comparison of knowledge scores between groups for sub-domains of short-term outcomes, long-term outcomes, numerical information, and treatments
Anxiety | within 24 hours of verbal counseling
  Comparison of change in participant anxiety as assessed by STAI

CONTACTS AND LOCATIONS:
Overall Officials: Mir A Basir, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert Hospital, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD.

REFERENCES:
- [Background] Cummings J; COMMITTEE ON FETUS AND NEWBORN. Antenatal Counseling Regarding Resuscitation and Intensive Care Before 25 Weeks of Gestation. Pediatrics. 2015 Sep;136(3):588-95. doi: 10.1542/peds.2015-2336. PMID 26324869
- [Background] Raju TNK, Mercer BM, Burchfield DJ, Joseph GF Jr. Periviable birth: executive summary of a joint workshop by the Eunice Kennedy Shriver National Institute of Child Health and Human Development, Society for Maternal-Fetal Medicine, American Academy of Pediatrics, and American College of Obstetricians and Gynecologists. Obstet Gynecol. 2014 May;123(5):1083-1096. doi: 10.1097/AOG.0000000000000243. PMID 24785861
- [Background] Muthusamy AD, Leuthner S, Gaebler-Uhing C, Hoffmann RG, Li SH, Basir MA. Supplemental written information improves prenatal counseling: a randomized trial. Pediatrics. 2012 May;129(5):e1269-74. doi: 10.1542/peds.2011-1702. Epub 2012 Apr 9. PMID 22492766
- [Background] Paivio A. Dual coding theory: Retrospect and current status. Can J Psychol. 45(3):255-87, 1991
- [Derived] Rau NM, Mcintosh JJ, Flynn KE, Szabo A, Ahamed SI, Asan O, Hasan MK, Basir MA. Multimedia tablet or paper handout to supplement counseling during preterm birth hospitalization: a randomized controlled trial. Am J Obstet Gynecol MFM. 2023 Apr;5(4):100875. doi: 10.1016/j.ajogmf.2023.100875. Epub 2023 Jan 26. PMID 36708966